CLINICAL TRIAL: NCT06112795
Title: Exploring Cultural Acceptability of Community Breast Cancer Risk Assessment Among Hispanic Women in Maricopa County
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-001884; NCI-2023-00465 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-001884 (Other: Mayo Clinic in Arizona)
Record Dates: First submitted 2023-09-27; First posted 2023-11-01 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Breast Carcinoma; Breast Cancer; Breast Cancer Female
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Participants attend an interview or participate in a focus group on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study explores the cultural acceptability of community breast cancer risk assessment among Hispanic women in Maricopa county.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the association between perceived risk and mammography screening behavior and differences in perceived risk by patient characteristics in Hispanic women screened at Mountain Park Health Center (MPHC).

II. Characterize attitudes, beliefs, and barriers towards mammography screening and cultural acceptability of BRCA models in community settings using focus group and interview data from under- and uninsured Hispanic women in Maricopa County.

OUTLINE: This is an observational study.

Participants attend an interview or participate in a focus group on study.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1:

  * Completed a baseline survey for the Latinas Learning about Density (LLEAD) study
  * Self-identify as Hispanic
  * Between 40-65 years of age
* AIM 2:

  * Between the ages of 45 and 65
  * Self-identify as Hispanic
  * Current residence in Maricopa County
  * Be under- (e.g. Arizona Health Care Cost Containment System) or uninsured at the time of enrollment
  * Can read and speak English or Spanish well enough to understand and complete the informed consent process and take part in either a focus group or individual interview

Exclusion Criteria:

* AIM I:

  * Women with a history of breast cancer
* AIM 2:

  * Women with a history of breast cancer

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Under and uninsured Hispanic women living in Maricopa county
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Mammography screening behavior | Baseline (at enrollment)
  Mammography screening behavior will be measured using two self-reported items: 1) history of ever having a mammogram, with a yes/no response and 2) history of last (most recent) mammogram" with the following response options: within the past year; at least 1, but less than 2 years ago; at least 2, but less than 5 years ago; 5 or more years ago; don't remember. Using these two items, a new variable of mammography screening behavior will be created, defined as the number of prior mammograms, categorizing responses as 0, 1 to 2, and 2+.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica D. Austin, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials